CLINICAL TRIAL: NCT04866407
Title: Essential Oils and Delayed Onset Muscle Soreness; The Effects of Topical Mentha x Piperita and Eucalyptus Globulus Oils in the Older Adult and Elderly Population
Brief Title: Topical Eucalyptus Globulus and Mentha x Piperita on Muscle Soreness in Older Adults and the Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sydney Asselstine, MD, Resident Physician, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021000112
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-06

CONDITIONS: Muscle Soreness
Keywords: Essential Oils; Muscle Soreness; Mentha x piperita; Eucalyptus globulus
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mentha x piperita (Experimental): A diluted solution of Mentha x piperita in carrier oil will be applied to the subject's interventional extremity.
  Interventions: Other: Mentha x piperita
- Eucalyptus globulus (Experimental): A diluted solution of Eucalyptus globulus in carrier oil will be applied to the subject's interventional extremity.
  Interventions: Other: Eucalyptus globulus
- No intervention (No Intervention): Each participant will have one extremity that receives no essential oil intervention.

INTERVENTIONS:
Other: Mentha x piperita — 2% solution of Mentha x piperita diluted in fractionated coconut oil for topical application will be applied to one extremity of the subjects in the 'Mentha x piperita' group.
  Arms: Mentha x piperita
Other: Eucalyptus globulus — 2% solution of Eucalyptus globulus diluted in fractionated coconut oil for topical application will be applied to one extremity of the subjects in the 'Eucalyptus globulus' group.
  Arms: Eucalyptus globulus

SUMMARY:
Subjects over age 50 with no previous resistance training sessions will be recruited at a subacute rehabilitation and long term care facility.

Subjects will be asked to perform a series of eccentric upper arm curl exercises under physician supervision in order to induce muscle soreness. Afterwards, topical oil containing a 2% dilution of either eucalyptus or peppermint oil in fractionated coconut oil will be applied to the flexor surface of the proximal non-dominent arm, and plain fractionated coconut oil to the other arm. This will be repeated at 8 hours and 24 hours after exercise. Subjects will be asked to report their perceived level of muscle soreness using a visual analog scale survey 24, 48, and 72 hours after exercise.

DETAILED DESCRIPTION:
Subjects 50 years old and above with no previous resistance training sessions within the past year will be recruited at a subacute rehabilitation and long-term care facility. A verbal explanation will be provided to the potential subjects by investigators on-site at the facility, including the fact that their care at the facility will not be affected by their decision to participate or not, and if they are interested in proceeding they will be asked to complete a survey regarding the subject's demographics (gender, age, hand dominance) and medical history, ensure there are no hypersensitivities to the oils being used, upper extremity injuries within 1 year, and that they have the functional capacity for exercise of 3.5METs or greater based on the Duke Activity Status Index. If participants pass the screening process they will again be informed of the study and all potential risks/benefits prior to signing an informed consent.

Eucalyptus globulus and Mentha x piperita essential oils will be obtained commercially from SunRose Aromatics (Morrill, Maine), and, individually, will be mixed with carrier oil for application. SunRose Aromatics is a recommended supplier from the RJ Buckle Clinical Aromatherapy for Health Professionals course. Fractionated coconut oil will be used as the carrier oil and also obtained from SunRose Aromatics. A 2% oil mixture for topical application will be made with essential oils diluted in fractionated coconut oil per guidelines from the RJ Buckle Clinical Aromatherapy for Health Professionals course recommendations. This mixture will be prepared directly before application of oils. The unmixed oils will be stored in a private room with no windows at room temperature at the Manor Health and Rehabilitation facility (689 W Main St, Freehold, NJ 07728).

Participants will be divided randomly into the Mentha x piperita or the Eucalyptus globulus group. A 2% oil mixture for topical application will be made with essential oils from SunRise Aromatics diluted in fractionated coconut oil per guidelines from the RJ Buckle Clinical Aromatherapy for Health Professionals course recommendations. Physician-supervised eccentric exercise of the elbow flexors will be performed based on an adaptation of the method described by Weber. Free weight dumbbells will provide resistance. The subject will be instructed to prolong the extension aspect of the curl to be five seconds long. They will repeat this motion for 10 or more repetitions until exhaustion, either due to the participant feeling they can no longer tolerate the five second eccentric aspect of the exercise or the investigator identifying that their form has faltered. If subjects reach exhaustion after the 10 repetitions minimum, they will rest for 1 minute. If they are unable to complete 10 repetitions at this weight, the resistance will be decreased to the next lowest weight and they will continue until exhaustion. This will continue until subjects reach exhaustion with the lowest resistance weight. Immediately following exercise, the participants will have the respective oil applied topically to their left upper extremity by the investigator. Their right upper extremity will serve as the control and no essential oil will be applied. Investigators will apply the oil without any use of massage technique and to only apply very superficial pressure. This application will be repeated 8 hours after exercise, when DOMS has been known to initiate, and at 24 hours after exercise, when DOMS may begin to peak.

Subject outcomes will be based on a self-reported visual analog scale, which has previously been shown to have validity in subjectively quantifying perceived muscle soreness and used in prior studies. These outcomes will be recorded by investigators for both the intervention and control upper extremity at 24, 48, and 72 hours post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 50 years or older with no previous resistance training sessions in the past year
* Duke Activity Screening Index functional capacity of at least 3.5 metabolic equivalents or greater
* currently admitted at the Manor Health and Rehabilitation

Exclusion Criteria:

* history of musculoskeletal injury or weight bearing restrictions to the upper extremities within the past year
* known adverse reaction or allergy to the essential oils or hypersensitivities to fragrances
* open upper extremity wounds or history of upper extremity skin grafts

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Khan, MD, Principal Investigator — Rutgers RWJMS Department of Family Medicine
Locations (1):
- The Manor Health and Rehabillitation - CentraState, Freehold, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Do not plan to.

REFERENCES:
- [Background] Meamarbashi A. Herbs and natural supplements in the prevention and treatment of delayed-onset muscle soreness. Avicenna J Phytomed. 2017 Jan-Feb;7(1):16-26. PMID 28265543
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Hanif, M., Nisar, S., Khan, G., Mushtaq, Z., Zubair, M. (2019) Essential Oils. Essential Oil Research. Springer, Cham. doi: 10.1007/978-3-030-16546-8_1
- [Background] Baser, K., and Buchbauer, G. (2009) Handbook of Essential Oils: Science, Technology, and Applications. CRC Press LLC.
- [Background] de Sousa AA, Soares PM, de Almeida AN, Maia AR, de Souza EP, Assreuy AM. Antispasmodic effect of Mentha piperita essential oil on tracheal smooth muscle of rats. J Ethnopharmacol. 2010 Jul 20;130(2):433-6. doi: 10.1016/j.jep.2010.05.012. Epub 2010 May 19. PMID 20488237
- [Background] Kehili, S. et. al. Peppermint (Mentha piperita L.) essential oil as a potent anti-inflammatory, wound healing and anti-nociceptive drug. European Journal of Biological Research. 2020; 10(2):132-149. Doi: 10.5281/zenodo.3831042
- [Background] Vuong QV, Chalmers AC, Jyoti Bhuyan D, Bowyer MC, Scarlett CJ. Botanical, Phytochemical, and Anticancer Properties of the Eucalyptus Species. Chem Biodivers. 2015 Jun;12(6):907-24. doi: 10.1002/cbdv.201400327. PMID 26080737
- [Background] Liapi C, Anifandis G, Chinou I, Kourounakis AP, Theodosopoulos S, Galanopoulou P. Antinociceptive properties of 1,8-Cineole and beta-pinene, from the essential oil of Eucalyptus camaldulensis leaves, in rodents. Planta Med. 2007 Oct;73(12):1247-54. doi: 10.1055/s-2007-990224. Epub 2007 Sep 24. PMID 17893834
- [Background] Mascolo, N. et al. Biological screening of Italian Medicinal Plants for anti-inflammatory activity. Phytother Res. 1987; 1(1)28-31. Doi: 10.1002/ptr.2650010107
- [Background] Jun YS, Kang P, Min SS, Lee JM, Kim HK, Seol GH. Effect of eucalyptus oil inhalation on pain and inflammatory responses after total knee replacement: a randomized clinical trial. Evid Based Complement Alternat Med. 2013;2013:502727. doi: 10.1155/2013/502727. Epub 2013 Jun 18. PMID 23853660
- [Background] Gobel H, Schmidt G, Soyka D. Effect of peppermint and eucalyptus oil preparations on neurophysiological and experimental algesimetric headache parameters. Cephalalgia. 1994 Jun;14(3):228-34; discussion 182. doi: 10.1046/j.1468-2982.1994.014003228.x. PMID 7954745
- [Background] Gobel H, Schmidt G, Dworschak M, Stolze H, Heuss D. Essential plant oils and headache mechanisms. Phytomedicine. 1995 Oct;2(2):93-102. doi: 10.1016/S0944-7113(11)80053-X. PMID 23196150
- [Background] Weber MD, Servedio FJ, Woodall WR. The effects of three modalities on delayed onset muscle soreness. J Orthop Sports Phys Ther. 1994 Nov;20(5):236-42. doi: 10.2519/jospt.1994.20.5.236. PMID 7827630
- [Background] Zainuddin Z, Newton M, Sacco P, Nosaka K. Effects of massage on delayed-onset muscle soreness, swelling, and recovery of muscle function. J Athl Train. 2005 Jul-Sep;40(3):174-80. PMID 16284637
- [Background] Rey E, Lago-Penas C, Lago-Ballesteros J, Casais L. The effect of recovery strategies on contractile properties using tensiomyography and perceived muscle soreness in professional soccer players. J Strength Cond Res. 2012 Nov;26(11):3081-8. doi: 10.1519/JSC.0b013e3182470d33. PMID 22210472
- [Background] Tisserand, R., Young, R., & Williamson, E. M. (2014). The Skin. In Essential oil safety: A guide for health care professionals (pp. 69-98). Edinburgh: Churchill Livingstone/Elsevier
- [Background] Tisserand, R., Young, R., & Williamson, E. M. (2014). Essential Oil Profiles: Eucalyptus globulus. In Essential oil safety: A guide for health care professionals Edinburgh: Churchill Livingstone/Elsevier.
- [Background] Tisserand, R., Young, R., & Williamson, E. M. (2014). Essential Oil Profiles: Mentha x piperita. In Essential oil safety: A guide for health care professionals (pp. 69-98). Edinburgh: Churchill Livingstone/Elsevier. (pp. 387-391)
- [Background] Ainsworth BE, Haskell WL, Herrmann SD, Meckes N, Bassett DR Jr, Tudor-Locke C, Greer JL, Vezina J, Whitt-Glover MC, Leon AS. 2011 Compendium of Physical Activities: a second update of codes and MET values. Med Sci Sports Exerc. 2011 Aug;43(8):1575-81. doi: 10.1249/MSS.0b013e31821ece12. PMID 21681120

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mentha x Piperita | Eucalyptus Globulus
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mentha x Piperita | Eucalyptus Globulus | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 74 [64 to 84] | 72 [68 to 74] | 73 [64 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Perceived Muscle Soreness
Description: Perceived soreness using a visual analog scale rating from '0' to '100'; a higher score indicates more muscle soreness
Time Frame: 24 hours after exercise
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Mentha x Piperita | Eucalyptus Globulus
Number analyzed (Participants) | 4 | 4
score on a scale | 0 [0 to 0] | 14.58 [0 to 52]

2. Primary Outcome: Perceived Muscle Soreness
Description: Perceived soreness using a visual analog scale rating from '0' to '100'; a higher score indicates more muscle soreness
Time Frame: 48 hours after exercise
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Mentha x Piperita | Eucalyptus Globulus
Number analyzed (Participants) | 4 | 4
score on a scale | 17.6 [0 to 68] | 1.62 [0 to 4]

3. Primary Outcome: Perceived Muscle Soreness
Description: Perceived soreness using a visual analog scale rating from '0' to '100'; a higher score indicates more muscle soreness
Time Frame: 72 hours after exercise
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Mentha x Piperita | Eucalyptus Globulus
Number analyzed (Participants) | 4 | 4
score on a scale | 9.2 [0 to 37] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | Mentha x Piperita | Eucalyptus Globulus
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT04866407/Prot_SAP_000.pdf